CLINICAL TRIAL: NCT04559087
Title: Comparison of NOSES and Conventional Laparoscopic Surgery in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Xu Fujian, Xu Fujian, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA2020RW12
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Cancer
Keywords: Minimally invasive surgery; natural orififice specimen; radical resectiong of rectal cancer; laparoscopic surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Orifice Specimen Extraction Surgery (Experimental)
  Interventions: Procedure: Laparoscopic Surgery
- Conventional laparoscopy (Sham Comparator)
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Laparoscopic Surgery — NOSES:Natural orifice specimen extraction (NOSE) is the opening of a hollow viscus that already communicates with the outside world, such as the vagina or distal gastrointestinal tract, in order to remove a specimen. The premise of this technique is to reduce the trauma required to remove the specimen with the expectation that this may improve outcomes.
  Conventional Laparoscopic Surgery:Surgical specimens were taken out through abdominal wall.
  Other Names: Conventional Laparoscopic Surgery

SUMMARY:
Radical surgery for rectal cancer has evolved from the initial concept of total mesorctal excision (TME) to the wide application of laparoscopic surgery in the radical treatment of rectal cancer. After 30 years' rapid development, nowdays laparoscopic TME surgery for rectal cancer has become the first choice for those patients with rectal cancer. However, the auxiliary incision of the abdominal wall which is used to remove tumor specimens is contrary to the current concept of minimally invasive surgery. Avoiding abdominal wall incisions has become a common appeal of gastrointestinal surgeons and patients with rectal cancer. Natural orififice specimen extraction surgery (NOSES) can solve the problem of abdominal wall auxiliary incision, which complete rectal cancer radical resection and gastrointestinal reconstruction under the full laparoscopic. The specimens are taken out through the natural orifice (rectum or vagina) without an auxiliary incision, which is more in line with minimally invasive practice and easier to operate. Researching on the progress of laparoscopic radical resection of rectal cancer in NOSES aims to provide a certain reference for this operation.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were as follows: (1) patients aged between 18 and 80 years; (2) histopathology confirmed as colorectal adenocarcinoma; (3) preoperative imaging (CT and MR) assessments showed that colorectal cancer did not penetrate the serosa (≤T3); (4) tumor circumference <5 cm; (5) enhanced chest and abdominal pelvic CT scans before operation excluded liver metastasis, lung metastasis, and other distant organ metastases.

Exclusion Criteria:

* The preoperative exclusion criteria were as follows: (1) tumors could be resected by endoscopic submucosal dissection (ESD) and endoscopic mucosal resection (EMR); (2) body mass index (BMI) > 30 kg/m2; (3) patients with severe perforation, bleeding, or obstruction requiring emergency surgery; (4) recurrent cases; (5) patients undergoing neoadjuvant therapy or preoperative radiotherapy; (6) Anesthesiologists (ASA) score ≥ IV; (7) active period of infection; (8) blood neutrophils <3 × 109/L.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | One month after operation
  pulmonary infection，Urinary tract infection，anal function，intestinal obstruction，Anastomotic bleeding，etc.

SECONDARY OUTCOMES:
survival | 3-year and 5-year after operation
  3-year and 5-year Overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No